CLINICAL TRIAL: NCT06221124
Title: Ring-type Pulse Oximeter for Evaluation for Sleep Assessment Study
Acronym: ROSA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Belun Technology Company Limited (Other)
Collaborators: Stanford University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: SPO#179613
Record Dates: First submitted 2024-01-12; First posted 2024-01-24 (Actual); Last update posted 2024-01-24 (Actual); Status verified 2024-01

CONDITIONS: Sleep-Disordered Breathing; Sleep Architecture
MeSH Terms: conditions — Sleep Apnea Syndromes

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- BEL-Participant (Experimental): First, we will measure the size of the finger of the participant and select appropriate size of Belun Ring device and the participant will be instructed to wear it on a finger in addition to regular PSG set up on the night of sleep study. Simultaneous recording of Belun Ring data {pulse oximeter, pulse rate and actigraphy} and standard PSG will be performed for one night.
  Interventions: Device: Belun Ring Pulse Oximeter

INTERVENTIONS:
Device: Belun Ring Pulse Oximeter — Belun Ring Pulse Oximeter allows measurement and analysis of oximetry, pulse rate, photo-plethysmography (PPG), and accelerometer signals from the proximal phalanx of index finger. Sleep stage (bSTAGES) and respiratory event index (bAHI) are estimated.

SUMMARY:
Recently, various electronic lifestyle activity monitoring devices (ELAM) are increasingly commercially available. However, the quality and reliability of the data from ELAM are unclear, compared with polysomnography (PSG), which is the gold-standard sleep assessment method. Thus, combining ELAM with PSG will validate ELAM and improve its clinical and research utilization.

The investigators propose to conduct this study to validate ELAM device for sleep assessment. The investigators will compare Belun Ring data collection and overnight in-lab PSG measures of Sleep-Disordered Breathing (SDB) and sleep architecture in adults with obstructive sleep apnea (OSA) symptoms.

The investigators propose to recruit a total of 40 participants with symptoms of OSA. The overall accuracy, sensitivity and specificity of Belun Ring to assess SDB and sleep architecture will be validated by using PSG analysis as a gold standard.

ELIGIBILITY:
Inclusion Criteria:

* Age between 18 to 80 years old. Ideally balanced for sex and age (18 to 80 years old)
* no more than 75% of subjects in one bin of: (male, female)
* no more than 50% of subjects in one age-group (18-29, 30-39, 40-49, 50-59, 60-80)
* Patients with OSA symptoms (snoring, excessive daytime sleepiness or witnessed apnea, etc.)
* Without any unstable medical or psychiatric co-morbidities that would be expected to interfere with the study.
* If taking any medication, must be on a stable dose of medication for a month
* Able to read and understand English

Exclusion Criteria:

* Presence of any significant systemic or unstable medical condition which could lead to difficulty complying with the protocol, suicidality, current regular use of psychiatric medications, opiates, or thyroid medications, dementia, current substance abuse, post-traumatic or psychotic disorders, bipolar disorder; any significant neurologic disease, including possible and probable dementia, Parkinson's or Huntington's disease, brain tumor, progressive supranuclear palsy, seizure disorder, subdural hematoma, multiple sclerosis, history of significant head trauma, history of alcohol or substance use disorder within the past 2 years (DSM V criteria);
* If positive airway pressure (PAP) titration study or split night study (diagnostic and PAP titration study combined)

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2020-07-15 (Actual); Primary Completion 2021-12-01 (Actual); Study Completion 2023-06-12 (Actual)

PRIMARY OUTCOMES:
Validation with gold-standard polysomnography (PSG) recording | 1 year
  Concordance rate of bAHI from Belun Ring and apnea-hypopnea Index (AHI) from PSG

CONTACTS AND LOCATIONS:
Locations (1):
- Stanford Sleep Medecine Center, Redwood City, California, United States

IPD SHARING:
Plan to Share IPD: No